CLINICAL TRIAL: NCT02813005
Title: High Frequency Jet Ventilation for Percutaneous Interventional Radiology
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 6370
Record Dates: First submitted 2016-06-14; First posted 2016-06-24 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2016-06

CONDITIONS: Percutaneous Tumor Ablation
Keywords: High frequency jet ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Jet ventilation/ group A (Experimental): Frequency : 120-200/min Pressure : 1-2 bars Inspiratory fraction of oxygen : 100% and 50% if Expiratory pressure : 5 -10 cmH2O
  Interventions: Procedure: Jet ventilation group
- Standard ventilation/ group B (Sham Comparator): Apnea made by the anesthesiologist to the request of the radiologist.
  Interventions: Procedure: Standard ventilation group

INTERVENTIONS:
Procedure: Jet ventilation group — MONSOON III™ (Acutronic Medical System AG®, SEBAC) with Double lumen catheter 12CH (Acutronic Medical System AG®, SEBAC)
  Other Names: Frequence: 120-200/min; Pressure: 1-2 bars; Inspiratory fraction of Oxgen: 50%; Expiratory pressure: 5-10 cmH2O
  Arms: Jet ventilation/ group A
Procedure: Standard ventilation group — apnea made by the anesthesiologist to the request of the radiologist
  Other Names: apnea made by the anesthesiologist with Primus DRAGER Medical
  Arms: Standard ventilation/ group B

SUMMARY:
Evaluate benefits of High Frequency Jet Ventilation compare to standard ventilation during general anesthesia in patient undergoing peri diaphragmatic percutaneous tumor ablation.

The investigators hypothesis that procedure is shorter and more accurate in High Frequency Jet Ventilation group reducing target movement induced by ventilation.

ELIGIBILITY:
Inclusion Criteria:

* use of percutaneous ablation tumor techniques (<3cm) for inferior lung, superior kidney, superior liver or adrenal gland lesion

Exclusion Criteria:

* Severe chronic obstructive pulmonary disease
* Recent pneumothorax (one month)
* Recent thoracic surgery (one month)
* Body Mass Index > 40

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Time to hit the target | during the procedure
  Estimated the time for a puncture needle under High Frequency Jet Ventilation compared to the conventional mode of mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Sandra PETIOT, MD, Principal Investigator — Les Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaires de Starsbourg, Strasbourg, France